CLINICAL TRIAL: NCT01404923
Title: Assessment of On-demand MeteoSpasmyl® Use Effectiveness in Irritable Bowel Syndrome
Brief Title: Effectiveness of On-demand Meteospasmyl® Use in Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoires Mayoly Spindler (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMTO901
Record Dates: First submitted 2011-07-27; First posted 2011-07-28 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — alverine; Simethicone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- meteospasmyl (Experimental)
  Interventions: Drug: alverine citrate, simeticone
- standard of care (Active Comparator)
  Interventions: Drug: anti spasmodic agents

INTERVENTIONS:
Drug: anti spasmodic agents — best standard of care prescriptions
  Arms: standard of care
Drug: alverine citrate, simeticone — on-demand therapy
  Arms: meteospasmyl

SUMMARY:
The purpose of this study is to compare the effectiveness of 2 IBS treatment strategies:

* Strategy A = MeteoSpasmyl®, on-demand therapy
* Strategy B = standard of care chosen by the physician

ELIGIBILITY:
Inclusion Criteria:

* male or female ambulatory patients, aged >= 18 years
* with IBS as defined by Rome III criteria for more than 1 year and less than 10 years
* with a IBS-SSS between 175 and 400

Exclusion Criteria:

* Acute diarrhea, bowel disorders due to an underlying cause
* Patient treated with MeteoSpasmyl® within the past 6 months
* Recent history of gastro intestinal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2009-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

REFERENCES:
- [Result] Ducrotte P, Grimaud JC, Dapoigny M, Personnic S, O'Mahony V, Andro-Delestrain MC. On-demand treatment with alverine citrate/simeticone compared with standard treatments for irritable bowel syndrome: results of a randomised pragmatic study. Int J Clin Pract. 2014 Feb;68(2):245-54. doi: 10.1111/ijcp.12333. Epub 2013 Oct 21. PMID 24147869

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Meteospasmyl | Standard of Care
Started | 222 | 214
Completed | 199 | 197
Not Completed | 23 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Meteospasmyl | Standard of Care | Total
Number analyzed (Participants) | 222 | 214 | 436
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (14.9) | 55.1 (16.2) | 54.4 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 160 | 320
  Male | 62 | 54 | 116
Region of Enrollment [Number; unit: participants]
  France | 222 | 214 | 436

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Irritable Bowel Syndrome Quality Of Life Overall Score
Description: Irritable Bowel Syndrome Quality of Life total score (IBSQoL) is a health-related Quality of Life (QoL) disease-specific scale adapted for French patients. Total score ranges from minimum=0 to maximum = 100 representing the best outcome.
Time Frame: Baseline and 6 months
Population: The efficacy population included all patients with a calculable IBSQoL score at baseline and at least one of the following visit, i.e 173 and 167 patients, respectively in Meteospasmyl and standard of care group.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meteospasmyl | Standard of Care
Number analyzed (Participants) | 173 | 167
units on a scale | 13.8 (1.1) | 8.4 (1.2)
Statistical Analysis 1: Comparison: Meteospasmyl vs Standard of Care; Test type: Superiority or Other; p = 0.0008, ANCOVA; Mean Difference (Final Values) = 5.4

2. Primary Outcome: Percentage of Improvement of the Total IBSQoL Scores
Description: Improvement of the total IBSQoL scores from baseline to month 6 calculated in percentage
Time Frame: Baseline and 6 Months
Population: The efficacy population included all patients with a calculable IBSQoL score at baseline and at lesat one of the following visit, i.e 173 and 167 patients, respectively in Meteospasmyl and standard of care group.
Measure: Mean (Standard Deviation); unit: % of improvement of IBSQoL total scores
Arm/Group | Meteospasmyl | Standard of Care
Number analyzed (Participants) | 173 | 167
% of improvement of IBSQoL total scores | 28.5 (49.1) | 18.6 (37.2)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Four patients in standard of care group were excluded because no data available (Lost of follow up)
Arm/Group | Meteospasmyl | Standard of Care
Serious Adverse Events (participants affected / at risk) | 5/222 | 1/210
Other Adverse Events (participants affected / at risk) | 5/222 | 0/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Meteospasmyl (N=222) | Standard of Care (N=210)
pyloroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) — pre-existing disabling disorders of gastric emptying requiring surgery. Unexpected and not related to study drug.
transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) — Pre-existing hypertension and diabetes.Unexpected and not related to study drug
Sigmoiditis abcess intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) — sigmoid diverticulitis abscess. Unexpected, not related to study drug.
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Cancer of the cervix. Unexpected, not related to study drug
Electrical cardioversion (Surgical and medical procedures) | 1 (1) | 0 (0) — Medical history of hypertension, atrial fibrillation. Unexpected not related.
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Kidney tumor. Unexpected, not related.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Meteospasmyl (N=222) | Standard of Care (N=210)
Nausea, diarrhea, heartburn (Gastrointestinal disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days